CLINICAL TRIAL: NCT00557661
Title: A Multi-Center, Ascending Dose Trial to Assess the Safety, Pharmacokinetics and Pharmacodynamics of CD-NP Infusions in Patients With Congestive Heart Failure
Brief Title: Safety Study of CD-NP in Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nile Therapeutics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIL-CDNP-CT002
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Congestive Heart Failure
Keywords: Heart failure; CD-NP
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CD-NP — 24 hr intravenous infusion

SUMMARY:
An open-label study designed to determine the safety, tolerability and pharmacodynamics of CD-NP infusions in heart failure patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female ≥18 years of age diagnosed with NYHA class III or IV heart failure in the last six months
* Female patients must be post-menopausal or surgically sterile
* Diagnosed heart failure with left ventricular ejection fraction <40% obtained within the prior 6 months with at least one symptoms or signs of volume overload

Key Exclusion Criteria:

* Women who are pregnant, breast-feeding or of child-bearing potential
* Clinically unstable patients
* Major surgical procedures within 30 days of entry
* Febrile temp > 100 degrees F)
* Symptomatic carotid disease, critical carotid stenosis, or stroke within 3 months prior to study entry
* Currently on IV vasoactive support (e.g., heart transplant candidate)
* History of unexplained syncope within the past 3 months
* History of organ transplantation
* Comorbidities such as clinically significant cardiac valvular stenosis, aortic valvular disease, restrictive cardiomyopathy, hypertrophic obstructive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, infiltrative disease, uncorrected congenital heart disease, acute coronary syndrome, restrictive heart failure, or any other condition which, in the opinion of the Investigator, would prevent a patient's participation in the study.
* Participation in a clinical trial of any investigational therapy or device within 30 days prior to randomization.
* Treatment with nesiritide within 14 days prior to dosing.
* Inability to effectively communicate with study personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of CD-NP infusions in patients with heart failure | 28 days

SECONDARY OUTCOMES:
To evaluate the effect of CD-NP infusions on urinary flow rate, urinary sodium and potassium excretion | 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Steven Goldsmith, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis